CLINICAL TRIAL: NCT07291141
Title: A Comparative Study of MRI and Ultrasound for Detection of Primary Hepatocellular Carcinoma, Body Composition and Risk Factors for Decompensation in Liver Cirrhosis
Acronym: DETECT-HCC
Status: Recruiting | Type: Observational
Sponsor: Mattias Ekstedt (Other Government)
Collaborators: Antaros Medical (Industry); Amra Medical AB (Industry); Region Östergötland (Other); Region Jönköping County (Other Government); Västra Götalandsregionen (Other); Region Stockholm (Other Government); Örebro County Council (Other Government); Uppsala County Council, Sweden (Other Government); Norrlands Universitetssjukhus, Umea, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Mattias Ekstedt, Consultant/Senior associate professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Other Study IDs: 2024-02472-01; CIV-23-08-043855 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhoses; Hepatocellular Carcinoma (HCC); Sarcopenia in Liver Cirrhosis; Portal Hypertension Related to Cirrhosis; MRI; Ultrasound
Keywords: Abbreviated MRI; Hepatocellular carcinoma; Liver cirrhosis; Sarcopenia
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, whole blood, liver biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with liver cirrhosis without prior hepatocellular carcinoma

SUMMARY:
DETECT-HCC-ESLD is a prospective multicenter study designed to examine early detection and risk stratification of hepatocellular carcinoma (HCC) in individuals with advanced liver disease. Adults with cirrhosis of different etiologies are enrolled and followed longitudinally with structured clinical assessments and imaging at predefined intervals.

A key objective is to evaluate ultrasound and abbreviated MRI (AMRI) as surveillance modalities for HCC. The study examines detection performance, feasibility, and factors influencing image quality and interpretability.

The protocol also includes the study of body composition, focusing on how variations in adiposity and muscle mass may relate to imaging characteristics, disease progression, and HCC risk.

Longitudinal clinical and imaging data are used to explore prediction models aimed at identifying patients with differing levels of HCC risk. The study records outcomes such as incident HCC, liver-related complications, and mortality to support analyses of disease trajectories.

The DETECT-HCC-ESLD study provides a structured framework for collecting clinical, imaging, and body composition data over time, enabling detailed evaluation of surveillance strategies and risk patterns in advanced liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis, according to clinical practice. Based on criteria such as elastography, symptoms, biopsy, or radiology.
* Age ≥18 years ≤ 84
* Written informed consent from the participant

Exclusion Criteria:

* Contraindications for MRI (ferrrous material, claustrophobia)
* Pregnancy
* Diagnosis of primary sclerosing cholangitis (PSC)
* Vascular liver disease
* Congenital liver fibrosis
* Previous diagnosis of hepatic carcinoma (HCC)
* Previous liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with liver cirrhosis without prior hepatocellular carcinoma or liver transplant.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Lesion at high risk for hepatocellular carcinoma (HCC) - (LI RADS 4-5) | Baseline visit
  A nodule on MRI classified as LI-RADS 4 or 5 according to the American College of Radiology (ACR) LI-RADS criteria.
Lesion at high risk for hepatocellular carcinoma (HCC) - (LI RADS 4-5) | Visit 2 (6 months)
  A nodule on MRI classified as LI-RADS 4 or 5 according to the American College of Radiology (ACR) LI-RADS criteria.
Lesion at high risk for hepatocellular carcinoma (HCC) - (LI RADS 4-5) | Visit 3 (12 months)
  A nodule on MRI classified as LI-RADS 4 or 5 according to the American College of Radiology (ACR) LI-RADS criteria.
Lesion at high risk for hepatocellular carcinoma (HCC) - (LI RADS 4-5) | Visit 4 (18 months)
  A nodule on MRI classified as LI-RADS 4 or 5 according to the American College of Radiology (ACR) LI-RADS criteria.
Lesion at high risk for hepatocellular carcinoma (HCC) - (US LI RADS 3) | Baseline visit
  A nodule on ultrasound classified as US LI-RADS 3 according to the American College of Radiology (ACR) LI-RADS criteria
Lesion at high risk for hepatocellular carcinoma (HCC) - (US LI RADS 3) | Visit 2 (6 months)
  A nodule on ultrasound classified as US LI-RADS 3 according to the American College of Radiology (ACR) LI-RADS criteria
Lesion at high risk for hepatocellular carcinoma (HCC) - (US LI RADS 3) | Visit 3 (12 months)
  A nodule on ultrasound classified as US LI-RADS 3 according to the American College of Radiology (ACR) LI-RADS criteria
Lesion at high risk for hepatocellular carcinoma (HCC) - (US LI RADS 3) | Visit 4 (18 months)
  A nodule on ultrasound classified as US LI-RADS 3 according to the American College of Radiology (ACR) LI-RADS criteria
The Muscle Assessment Score (MAsS) | Baseline visit
  The Muscle Assessment Score (MAsS) combines thigh muscle z-score and muscle fat infiltration to detect muscle composition phenotypes.
The Muscle Assessment Score (MAsS) | Visit 2 (12 months)
  The Muscle Assessment Score (MAsS) combines thigh muscle z-score and muscle fat infiltration to detect muscle composition phenotypes.
The Muscle Assessment Score (MAsS) | Visit 3 (12 months)
  The Muscle Assessment Score (MAsS) combines thigh muscle z-score and muscle fat infiltration to detect muscle composition phenotypes.
The Muscle Assessment Score (MAsS) | Visit 4 (18 months)
  The Muscle Assessment Score (MAsS) combines thigh muscle z-score and muscle fat infiltration to detect muscle composition phenotypes.
Liver associated clinical events (LACE) | From enrollment and six months after the last study visit (after a total of 24 months).
  Any of clinical ascites, variceal bleeding, hepatic encephalopathy west haven >= grade 2, hepatorenal syndrome, or hepatopulmonary syndrome.

SECONDARY OUTCOMES:
Hepatocellular carcinoma (HCC) | From enrollment and six months after last visit (a total of 24 months).
  HCC verified by pathology.
Treatment for hepatocellular carcinoma | From enrollment and six months after last visit (a total of 24 months).
  Treatment given to patients that develope HCC: ablation, resection, TACE, systemic treatment, or best supportive care.
Death | From enrollment and six months after last visit (a total of 24 months).
  All cause mortality
Liver stiffness (VCTE) | Baseline
  Liver stiffness measured with Fibroscan
Liver stiffness (VCTE) | Visit 2 (6 months)
  Liver stiffness measured with Fibroscan
Liver stiffness (VCTE) | Visit 3 (12 months)
  Liver stiffness measured with Fibroscan
Liver stiffness (VCTE) | Visit 4 (18 months)
  Liver stiffness measured with Fibroscan
Liver stiffness (MRE) | Baseline
  Liver stiffness measured with magnetic resonance elastography (MRE)
Liver stiffness (MRE) | Visit 2 (6 months)
  Liver stiffness measured with magnetic resonance elastography (MRE)
Liver stiffness (MRE) | Visit 3 (12 months)
  Liver stiffness measured with magnetic resonance elastography (MRE)
Liver stiffness (MRE) | Visit 4 (18 months)
  Liver stiffness measured with magnetic resonance elastography (MRE)
Liver volume | Baseline
  Liver volume measured with MRI
Liver volume | Visit 2 (6 months)
  Liver volume measured with MRI
Liver volume | Visit 3 (12 months)
  Liver volume measured with MRI
Liver volume | Visit 4 (18 months)
  Liver volume measured with MRI
Spleen volume | Baseline
  Spleen volume measured with MRI
Spleen volume | Visit 2 (6 months)
  Spleen volume measured with MRI
Spleen volume | Visit 3 (12 months)
  Spleen volume measured with MRI
Spleen volume | Visit 4 (18 months)
  Spleen volume measured with MRI

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ekstedt, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of gastroenterology and hepatology, University hospital in Linköping, Linköping, Select A State Or Province, Sweden

IPD SHARING:
Plan to Share IPD: Undecided